CLINICAL TRIAL: NCT04241757
Title: Electrocardiogram in General Practice : the EGG Study
Acronym: EGG
Status: Terminated | Type: Observational
Why Stopped: The EGG study is no longer in progress, as the association that carried it out (IRMG) has had to close due to the impact of the Covid crisis on continuing education.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association CNGE IRMG (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRBN432019/CHUSTE
Record Dates: First submitted 2019-11-18; First posted 2020-01-27 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Indication for ElectroCardioGram
Keywords: ElectroCardioGram; General practice; Diagnosis; Signs and symptoms; Feasibility studies
MeSH Terms: conditions — Disease; Signs and Symptoms | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with indication of ElectroCardioGram (ECG): Patient with indication of ElectroCardioGram (ECG) will be included. They will have a collection of results ElectroCardioGram (ECG).
  Interventions: Diagnostic Test: ElectroCardioGram (ECG)

INTERVENTIONS:
Diagnostic Test: ElectroCardioGram (ECG) — Collection of results ElectroCardioGram (ECG).

SUMMARY:
Existing resources to assist interpretation of ElectroCardioGram (ECG) in general practice provide specialized and comprehensive reading based on pathologies and ElectroCardioGram (ECG) signs rather than ElectroCardioGram (ECG) indications.

Describing practices in general medicine could help prioritize the relevance of clinical and ECG signs for the general practitioner, enabling to adjust the reading given the context.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the clinical signs and ElectroCardioGram (ECG) in situations indicating an ElectroCardioGram (ECG) in general practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient consulting one of the generalist practitioner investigators
* In doctor's office or at home, scheduled or not,
* During normal surgery hours or out-of-hours service,
* Whatever the reason for consultation,
* Aged 18 years or older,
* Having an indication of ElectroCardioGram (ECG) and/or request certificate of non-contra-indication to the practice of physical activity certificate of non-contra-indication to the practice of physical activity

Exclusion Criteria:

* ElectroCardioGram (ECG) not performed due to emergency context
* Patient with cognitive impairment who cannot give consent to participate in the study and / or patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with indication of ElectroCardioGram (ECG) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Description of clinical signs | day 0
  Prevalence of each clinical sign within each Electrocardiogram indication
Description of clinical signs ElectroCardioGram (ECG) sign | day 0
  Prevalence of each sign on the Electrocardiogram within each indication.

SECONDARY OUTCOMES:
Difficulties in carrying out the Electrocardiogram | Day 0
  Duration of the Electrocardiogram (minutes) Measured by average duration of the ECG, prevalence of the difficulties of realization and interpretation mentioned by the investigators.
Initial management types | Months 1
  Prevalence of initial management types (certificate, medication, addressing) at 1 month.
Diagnosis types | Months 1
  Prevalence of diagnosis types at 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Paul FRAPPE, MD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- Association CNGE IRMG, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No